CLINICAL TRIAL: NCT06092749
Title: Effectiveness of Transgrade vs Interlaminar Epidural Steroid Injection for Chronic Unilateral Lumbar Radicular Pain
Brief Title: Chronic Unilateral Lumbar Radicular Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ibrahim Mamdouh Esmat, Assistant Professor of Anesthesia, Intensive Care and Pain Management Department, Faculty of Medicine, Ain- shams University, Cairo, Egypt., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU MD 286/ 2023
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transgrade technique (TG) (Active Comparator)
  Interventions: Other: Transgrade technique (TG)
- Interlaminar technique (IL) (Active Comparator)
  Interventions: Other: Interlaminar technique (IL)

INTERVENTIONS:
Other: Transgrade technique (TG) — Transgrade (TG) Epidural Steroid Injection technique
  Arms: Transgrade technique (TG)
Other: Interlaminar technique (IL) — Interlaminar (IL) Epidural Steroid Injection technique
  Arms: Interlaminar technique (IL)

SUMMARY:
Chronic neuropathic lumbar pain is among one of the most widespread complaints of patients.Many approaches have been attempted to target chronic pain, with varying efficacy and risks. Transgrade (TG) epidural injection is a new technique using a Racz- Coudé needle for epidural access at a "transgrade" angle without requiring any specialized hardware or accessories. Interlaminar (IL) epidural steroid injection (ESI) is one of the procedures that involves the delivery of injectate to the epidural space through directing a needle between the laminae of two adjacent vertebrae.

ELIGIBILITY:
Inclusion Criteria:

* > 6-month history of persistent pain in one leg with back pain.
* Capable of giving informed consent.
* Unsatisfactory response to conventional treatments including physical therapy or medications with a numeric rating scale (NRS) ≥ 5.

Exclusion Criteria:

* Previous lumbar spinal surgery.
* Myelopathy.
* Rheumatoid disorders.
* Psychiatric disorders
* Bleeding or coagulation disorders

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
The average numeric rating scale (NRS) pain scores | at 12 weeks after intervention
  The numeric rating scale (NRS) is most commonly 0 to 10, with 0 being "no pain" and 10 being "the worst pain imaginable."

CONTACTS AND LOCATIONS:
Locations (1):
- Ain-Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No